CLINICAL TRIAL: NCT07173309
Title: Evaluation of Eye Gaze Sharing in the Operating Room
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nicholas Kavoussi, Assistant Professor Department of Urology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 231997B; 1R21EB035783-01 (NIH)
Record Dates: First submitted 2025-08-29; First posted 2025-09-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Kidney Stones
Keywords: Kidney Stones; Augmented Reality; Gaze Guidance
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR guided (Experimental): Trainees can see experts' gaze through the HoloLens
  Interventions: Device: Augmented reality
- Non-AR guided (No Intervention): Trainees cannot see experts' gaze through the HoloLens. This should be the standard of care control group.

INTERVENTIONS:
Device: Augmented reality — Augmented reality markers show the surgical trainee the expert's gaze location during the kidney exploration phase of surgery.
  Arms: AR guided

SUMMARY:
This project aims to develop an augmented reality (AR) tool to enhance skill acquisition for endoscopic kidney stone surgery. Of the 100,000 patients who undergo an endoscopic kidney stone treatment annually in the United States, 25% will require a repeat stone surgery within 20 months of their index surgery. The repeat stone surgery rate is almost completely driven by postoperative residual stone fragments, which lead to ureteral obstruction, causing pain, urinary tract infection, and kidney injury. One significant factor that contributes to residual stone fragments is limited visualization of the entire collecting system - a skill directly associated with surgeon experience. This leads to novice surgeons having a much higher recurrence rate than experienced ones. As the incidence of kidney stone disease continues to increase (prevalence of 10%, incidence of 1116 per 100,000), improved endoscopic surgical training is required to improve outcomes of stone surgeries and minimize complications by improving stone-free rate.

Currently, skill assessment during endoscopic stone surgery is limited. There are no objective metrics for endoscopic surgery to assess skill. The only feedback trainees get is in the form of verbal communication from expert surgeons, usually after the conclusion of surgery. Thus, most feedback is synoptic and limited in facilitating skill acquisition. Operative time and patient safety concerns restrict the amount of active, real-time feedback given during a case for skill acquisition. Endoscopic kidney stone surgery is uniquely challenging given the small depth and field of view of current endoscopes, which complicate the complete visualization of the entire collecting system.

Navigation of the collecting system relies on mentally mapping preoperative imaging to the endoscopic surgical field. Success in mapping relies on hand-eye coordination, memory, and spatial reasoning, which are gained through practice. Thus, there is a need for tools that facilitate endoscopic surgical skill acquisition.

The overarching hypothesis for this research is that surgical skill acquisition and outcomes for endoscopic kidney stone surgery can be improved by analyzing eye gaze data and using expert gaze to guide surgical trainees intraoperatively. Eye gaze guidance has been shown to lead to better skill acquisition in virtual reality surgical tasks compared with motion guidance alone. The proposed system would provide real-time education for trainees during endoscopic stone surgery, such as through head-mounted displays (i.e., the Microsoft HoloLens 2). The investigators have previously demonstrated eye gaze sharing in phantoms. By implementing this system in the operating room (OR), the investigators would be able to instill durable skill acquisition in trainees. The investigators will also implement the NASA-task load index for the trainees to gauge the usability of the system.

DETAILED DESCRIPTION:
Specifically for this study, the investigators are asking surgical trainees and experts to wear the HoloLens 2 in the operating room while conducting kidney stone surgery. The investigators measure the eye gaze data of the trainee and expert using the HoloLens. In the experimental arm of the trial, the trainees get visual guidance through a hologram showing the expert's gaze in addition to the verbal guidance as their standard of care. The intervention is only during the kidney exploration phase of the surgery. The augmented reality is turned off during the rest of the surgery, which proceeds per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Urology residents at Vanderbilt University Medical Center

Exclusion Criteria:

-

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Completeness of kidney exploration | 1-10 minutes
  Percentage of kidney that was visualized

SECONDARY OUTCOMES:
Gaze path of the user while performing kidney exploration | 1-10 minutes
  Extracted from eye-camera recording from the HoloLens 2

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the endoscope video and eye-gaze information from the study, and associated metadata, including the study protocol.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will be uploaded to the NIDDK repository by Aug 2026. We foresee the data being available indefinitely.
Access Criteria: Access to individual data will be controlled through the NIDDK repository and available only for research purposes.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT07173309/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT07173309/ICF_001.pdf